CLINICAL TRIAL: NCT00180804
Title: Combination of Maternal KIR and Fetal HLA-C Genes in Recurrent Miscarriages
Brief Title: Maternal KIR and Fetal HLA-C Genes in Recurrent Miscarriages
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 05/MRE02/20
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Recurrent Miscarriages
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
For implantation of developing conceptus, placental cells need to invade mother's uterus to access maternal blood supply in a control manner. We have found a combination of maternal immune genes (the KIR family) and fetal genes (HLA-C) strongly associated with pre-eclampsia where placenta does not implant adequately. The aim of this research is to investigate these two genes family in women suffering with recurrent miscarriages and find a possible link between them.

DETAILED DESCRIPTION:
Little is known about reasons for early pregnancy failures. It is believed that some pathology leading to defective implantation of fetus in maternal uterus may lead to recurrent early miscarriages. This project arises from previous work on pre-eclampsia where we found combination of maternal immune genes (KIR) with their ligand (HLA-C) in the fetus was strongly associated with the disease. We will tissue type the fetus, mother and father in cases of unexplained miscarriages. We hope that genetic findings in recurrent miscarriage will lead to new insights, prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

Couples with 3 or more unexplained miscarriages

Exclusion Criteria:

Previous livebirths, parental karyotypic abnormalities, thrombophilic defects, uterine structural abnormalities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-04; Study Completion 2005-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Moffett, MRCP, Principal Investigator — University of Cambridge, UK; Raj Rai, MRCOG, Principal Investigator — Imperial College London; Preeti Jindal, MRCOG, Principal Investigator — St. Mary's NHS Trust, London; Winnie Lo, Principal Investigator — St. Mary's NHS Trust, London
Locations (1):
- St. Mary's Hospital, London, United Kingdom